CLINICAL TRIAL: NCT05992337
Title: New Biomarkers in the Prediction of Chemotherapy-induced Cardiotoxicity.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiology Prague (Network)
Collaborators: BioVendor LM (Unknown); Oncology Center Medicon (Unknown)
Responsible Party: Sponsor
Other Study IDs: Version_Protocol_3_5_2021
Record Dates: First submitted 2021-09-28; First posted 2023-08-15 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Cardiotoxicity; Chemotherapy Effect; Chemotherapy Induced Systolic Dysfunction
MeSH Terms: conditions — Cardiotoxicity | interventions — Blood Specimen Collection; Echocardiography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with breast cancer treated with chemotherapeutics without signs of cardiotoxicity
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Echocardiography; Diagnostic Test: 24-hours monitoring of ECG
- Women with breast cancer treated with chemotherapeutics with signs of cardiotoxicity
  Interventions: Diagnostic Test: Blood sampling; Diagnostic Test: Echocardiography; Diagnostic Test: Cardio MRI; Diagnostic Test: 24-hours monitoring of ECG; Diagnostic Test: 24 hours monitoring of BP

INTERVENTIONS:
Diagnostic Test: Blood sampling — Blood sample collection for mRNA determination
Diagnostic Test: Echocardiography — Echocardiography for detection of ventricular dysfunction
Diagnostic Test: Cardio MRI — MRI for early detection of myocardial impairment caused by chemotherapy
  Groups: Women with breast cancer treated with chemotherapeutics with signs of cardiotoxicity
Diagnostic Test: 24-hours monitoring of ECG — Diagnostic test for detection of arrhythmias as a consequence of cardiotoxicity
Diagnostic Test: 24 hours monitoring of BP — Diagnostic test for detection of hypertension as a consequence of cardiotoxicity
  Groups: Women with breast cancer treated with chemotherapeutics with signs of cardiotoxicity

SUMMARY:
Early detection and thus rapid therapy of cardiotoxicity related to chemotherapy are essential for restoring cardiovascular function. The complete recovery of the cardiovascular system decreases with time to identify the presence of cardiotoxic damage. The project aims to define new biomarkers for the early detection of cardiotoxicity in patients treated with chemotherapy.

DETAILED DESCRIPTION:
The most effective approach to minimizing the consequences of cardiotoxicity of oncological treatment is its early identification, adjustment of oncological treatment (change of procedure, dose, drugs), and immediate initiation of cardiovascular therapy. However, the current standard for monitoring the cardiovascular system in cancer patients identifies cardiotoxicity only if functional impairment has already occurred, which precludes any chance of effective prevention. The aim of the project is to identify new biomarkers for the early detection of the cardiotoxic effect of chemotherapy in women with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer
* Chemotherapy with a known cardiotoxic side effect

Exclusion Criteria:

* Known cardiovascular disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast cancer chemotherapy population
Study Population: Women with breast cancer
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Early detection of the cardiotoxic effect of chemotherapy using new biomarkers | one year follow-up.
  Echocardiography and MRI detection of cardiotoxic effect of chemotherapy - dysfunction of left ventricle, arrythmias, hypertension

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Cardiology Prague Ltd, Prague
  - Oncology Center Medicon, Prague